CLINICAL TRIAL: NCT03481998
Title: A Phase IB/II to Evaluate Efficacy and Safety of SHR6390 in Combination With Letrozole or Anastrozole or Fulvestrant in Patients With HR Positive and HER2 Negative Recurrent/Metastatic Breast Cancer
Brief Title: A Study of SHR6390 in Combination With Letrozole or Anastrozole or Fulvestrant in Patients With HR Positive and HER2 Negative Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR6390-Ib/II-201
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Advanced Breast Cancer
Keywords: CDK4/6 inhibitor; Breast cancer; Postmenopausal women; Hormone-receptor positive; HER2 negative; Premenopausal women
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Part 1) (Experimental): Participants receive SHR6390 (at protocol defined dose levels) in combination with letrozole 2.5 mg or anastrozole 1mg, orally once daily (continuously).
  Interventions: Drug: SHR6390; Drug: Letrozole or anastrozole or Fulvestrant
- Cohort 2 (Part 1) (Experimental): SHR6390 (TBD), in combination with letrozole 2.5 mg or anastrozole 1mg, orally once daily (continuously).
  Interventions: Drug: SHR6390; Drug: Letrozole or anastrozole or Fulvestrant
- SHR6390 + Letrozole or anastrozole (Part 2) (Experimental): SHR6390 (RP2D, recommended Phase 2 dose), in combination with letrozole 2.5 mg or anastrozole 1mg, orally once daily (continuously).
  Interventions: Drug: SHR6390; Drug: Letrozole or anastrozole or Fulvestrant
- SHR6390 + Fulvestrant Cohort 3 (Part 1) (Experimental): SHR6390 (at protocol defined dose levels), in combination with Fulvestrant 500 mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 for every cycle once daily
  Interventions: Drug: SHR6390; Drug: Letrozole or anastrozole or Fulvestrant
- SHR6390 + Fulvestrant Cohort 4 (Part 1) (Experimental): SHR6390 (TBD), in combination with Fulvestrant 500 mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 for every cycle once daily
  Interventions: Drug: SHR6390; Drug: Letrozole or anastrozole or Fulvestrant

INTERVENTIONS:
Drug: SHR6390 — SHR6390 150 mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
Drug: Letrozole or anastrozole or Fulvestrant — Letrozole 2.5mg or anastrozole 1mg, orally once daily (continuously)， or Fulvestrant 500mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 for every cycle until progressive disease

SUMMARY:
This is a phase IB/II clinical trial to evaluate the efficacy and safety of SHR6390 in combination with Letrozole or Anastrozole or Fulvestrant. Patients who have HR positive and HER2 negative recurrent/metastatic breast cancer and have not received systemic anticancer therapy are eligible for study.

ELIGIBILITY:
Inclusion Criteria:

1. Has the pathologically-confirmed diagnosis of locally recurrent or metastatic, hormone-receptor positive, HER2 negative Breast Cancer.
2. Age: 18 - 75 years old, postmenopausal women.prepostmenopausal women, but should receive Ovary castration.

   Inclusion Criteria
3. Cohort 1 and Cohort 2 :No prior systemic anti-cancer therapy for advanced HR+ disease.

Cohort 3 and Cohort 4 : Patients must satisfy the following criteria for prior therapy:

1. a) Progressed after 2 years during treatment of adjuvant therapy with an aromatase inhibitor if postmenopausal, or tamoxifen if pre- or perimenopausal.

   b)Progressed within 12 months of completion of adjuvant therapy with an aromatase inhibitor if postmenopausal, or tamoxifen if pre- or perimenopausal.

   c) Progressed while 6 month after the end of prior aromatase inhibitor therapy for advanced/metastatic breast cancer if postmenopausal, or prior endocrine treatment for advanced/metastatic breast cancer if pre- or perimenopausal.
2. One previous line of chemotherapy for advanced/metastatic disease is allowed in addition to endocrine therapy.

4. Eastern Cooperative Oncology Group [ECOG] 0-1 Measurable disease as per Response Evaluation Criterion in Solid Tumors[RECIST] 1.1

5. Adequate organ and marrow function

Exclusion Criteria

1. Confirmed diagnosis of HER2 positive disease
2. Patients who received any endocrine therapy as neo/adjuvant therapy for breast cancer are eligible. If the neo/adjuvant therapy of any endocrine therapy , the disease-free interval must be greater than 12 months from the completion of treatment until study entry.
3. Patients who received prior treatment with any CDK4/6 inhibitor, everolimus,fulvestant.
4. Clinically significant cardiovascular and cerebrovascular diseases,including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), or ventricular arrhythmia which need medical intervention.
5. Has known active central nervous system metastases.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With adverse events (AEs) and serious adverse events (SAEs) at Phase 1 | Up to 4 weeks
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.
  Up to 24 months.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SHR6390 | Up to 4 weeks
Peak Plasma Concentration (Cmax) of SHR6390 | Up to 4 weeks
The time of SHR6390 to reach the maximum concentration (Tmax) | Up to 4 weeks
Half-time (t1/2) of SHR6390 | Up to 4 weeks
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to approximately 24 months.
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ¡Ý30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Progression-free Survival (PFS) per RECIST 1.1 | Up to approximately 24 months.
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) per RECIST 1.1 | Up to approximately 24 months.
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or SD per RECIST 1.1.
Number of Participants With adverse events (AEs) and serious adverse events (SAEs) | Up to approximately 24 months.
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Binhe Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - Ha'erbin Tumor Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Sir Run Run Shaw Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Q, Zhang P, Yan M, Yan X, Wang X, Gu Y, Qu X, Li S, Xu G, Zhu X, Xu B. Dalpiciclib in combination with letrozole/anastrozole or fulvestrant in HR-positive and HER2-negative advanced breast cancer: results from a phase Ib study. Ther Adv Med Oncol. 2024 Sep 2;16:17588359241273026. doi: 10.1177/17588359241273026. eCollection 2024. PMID 39229468